CLINICAL TRIAL: NCT03928366
Title: Synchronous Effect of Anesthetics on fMRI, EEG and Clinical Responses. Development of a More Precise System for Monitoring Anesthetic Effect.
Brief Title: Synchronous Effect of Anesthetics on fMRI, EEG and Clinical Responses
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Parc de Salut Mar (Other)
Responsible Party: Principal Investigator, Juan Luis Fernández Candil, PhD. Principal investigator., Parc de Salut Mar
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Basic Science
Other Study IDs: UNLOCK
Record Dates: First submitted 2019-04-11; First posted 2019-04-26 (Actual); Last update posted 2022-09-30 (Actual); Status verified 2022-09

CONDITIONS: Sedative Overdose
Keywords: Propofol, remifentanil, hypnosis, EEG, fMRI,
MeSH Terms: interventions — Propofol; Remifentanil

STUDY DESIGN:
Intervention Model Description: Volunteers receiving propofol and then remifentanil.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Volunteers receiving propofol and remifentanil (Experimental): Volunteers receive propofol to the loss of consciousness. Then they receive remifentanil during 12 min (pain stimuli in their finger also)
  Interventions: Drug: Propofol; Drug: Remifentanil

INTERVENTIONS:
Drug: Propofol — sedation
  Other Names: remifentanil
Drug: Remifentanil — remifentanil

SUMMARY:
Background: The mechanisms of action of intravenous anesthetics are unclear and the current monitors have limitations.

This signifies difficulties when assessing the correct dosage due to the considerable inter-individual variability of the patients, particularly in the elderly or seriously ill. It is necessary to customize the administration of anesthetics as underdosage can lead to the patient awareness during aggressive procedures, and over-dosage can cause serious complications and even augment mortality.

Objective: To design a new monitoring system of the levels of consciousness and analgesia in anesthetized subjects which is more accurate than those currently employed. It will be based on the synchronic changes of functional magnetic resonance (fMR) and electroencephalograph (EEG) readings, and clinical responses.

Methodology: Thirty healthy volunteers will be given propofol and remifentanil in different combinations, and painful stimuli will be also applied. The principal variable will be fMR images obtained by echo-planar imaging sequences. Real time will be correlated with cortical connectivity maps, EEG parameters (qCON, qNOX), clinical responses, and concentrations of anesthetics measured by pharmacokinetic and pharmacodynamic models (TCI).

DETAILED DESCRIPTION:
Main goal:

Develop a system for monitoring the effect of anesthetics on consciousness and pain, based on synchronous changes in functional neuroimaging, EEG and clinical responses.

Secondary objectives:

* Analyze the changes produced in the cortical connectivity map during the induction of anesthesia to understand the process of "advancement".
* Know more accurately the neuronal circuits involved in propofol-induced sleep.
* Study if the application of a known painful stimulus modifies in any way (clinical, EEG or by RMf) the LOC that has just been reached.
* Establish propofol dosing guidelines adjusted to each patient, studying if they reach the LOC at "sedative" or "hypnotic" doses.
* Establish remifentanil dosing guidelines, adjusted to each patient, studying the concentration of remifentanil to which the pain response in neuroimaging is inhibited (activation deactivation neuronal in fMRI).
* Validate existing mathematical models in relation to plasma and brain concentrations of propofol and remifentanil.
* Validate the value of clinical signs to predict whether a patient feels the painful stimulus received.

ELIGIBILITY:
Inclusion Criteria:

* Healthy adult volunteers (ASA 1 physical state) who agree to participate voluntarily in the study, previous information about it by the Principal Investigators (IP).

Exclusion Criteria:

* Psychological, psychiatric or neurological disorders. Consumption of drugs. Alterations cutaneous or anatomical cranial. Idiomatic or communication barrier. Allergy to propofol, remifentanil or to some of its excipients. Body mass index (BMI) <18 or> 30 kg / m2. Pregnancy. Airway or ventilation criteria hard. Absence of accompanying adult at the end of the study.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2017-06-13 (Actual); Primary Completion 2019-01-09 (Actual); Study Completion 2021-06-30 (Actual)

PRIMARY OUTCOMES:
Time and dose of propofol at loss of consciousness(LOC) | 10-15 min
  Volunteers stop tightening pneumatic pear. We register time and dose of propofol when the volunteer stops tightening pneumatic pear.
Register EEG and neuroimage during remifentanil administration. | 10-15 min
  After LOC, volunteers receive increasing doses of remifentanil and painful stimuli in the nail bed. If apnea, stop infusion remifentanil Volunteers receive increasing doses of remifentanil and painful stimuli in the nail bed. If apnea, stop infusion remifentanil. We registered time, dose, saturation and breathing frequency in every volunteer.

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital del Mar, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: Yes
Participants will be introduced to the fMRI The head will be set to try to prevent involuntary movements associated with the LOC. Routine by pulse oximetry, non-invasive blood pressure and electrocardiogram (ECG). It will be administered oxygen at 2 liters / min by nasal cannula with capnography line and transcutaneous carbon dioxide will be monitored. Volunteers will not be premedicated.
  EEG activity and fMRI images, as detailed in the section "Study variables". Each series of acquisitions will consist of a "resting state" (rs-fMRI), in which the subject will be asked to close their eyes and leave the mind ramble without further slogans, and also a series of tasks in which the participant will be exposed to a sequence of perceptive and nociceptive stimuli in order to objectify the effect of the drug on the nervous system central. The signal extracted from the RMf images will allow to study the dynamics of the metabolic changes and neurons in the brain with a temporal resolution.
Supporting Information: Study Protocol
Time Frame: 3 years
Access Criteria: volunteers without exclusion criteria

REFERENCES:
- [Background] Borrat X, Ubre M, Risco R, Gambus PL, Pedroso A, Iglesias A, Fernandez-Esparrach G, Gines A, Balust J, Martinez-Palli G. Computerized tests to evaluate recovery of cognitive function after deep sedation with propofol and remifentanil for colonoscopy. J Clin Monit Comput. 2019 Feb;33(1):107-113. doi: 10.1007/s10877-018-0134-3. Epub 2018 Mar 27. PMID 29589170